CLINICAL TRIAL: NCT04810052
Title: Feasibility of a Positive Activity Intervention in Cancer Patients From Collectivist Cultures
Brief Title: Positive Activities Intervention to Improve Quality of Life in Collectivist Culture Cancer Patients and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0789; NCI-2020-14194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0789 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-24; First posted 2021-03-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Behavior Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition I (contribution) (Experimental): Patients do 1 nice thing (can be as large or as small as they wish) BIW for 4 weeks for their caregivers while at home.
  Interventions: Behavioral: Behavioral Intervention; Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Condition II (gratitude) (Experimental): Patients write a letter or note of gratitude BIW for 4 weeks to their caregivers who have helped with their treatment or recovery.
  Interventions: Behavioral: Behavioral Intervention; Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Condition III (daily activities tracking) (Active Comparator): Participants keep track of their daily activities.
  Interventions: Behavioral: Behavioral Intervention; Other: Interview; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Perform 1 nice thing
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Condition I (contribution)
Behavioral: Behavioral Intervention — Write a letter or note of gratitude
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Condition II (gratitude)
Behavioral: Behavioral Intervention — Track daily activities
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Condition III (daily activities tracking)
Other: Interview — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the feasibility of two positive activities in improving quality of life in collectivist culture cancer patients and their caregivers. Cancer patients of collectivist cultures (e.g., Latinos, Asian Americans, African Americans) have been found to experience lower quality of life and more distress and depression when compared to those of individualist cultures, such as European Americans. Following a cancer diagnosis, collectivist patients may experience a change in their relationships with other family members and their roles within the family. The cancer diagnosis may lead to changes in roles and responsibilities, such as when a male breadwinner is no longer able to work due to hospital treatments. The two positive activities are designed to increase a sense of competence, autonomy, and connectedness, including contributing to household responsibilities (an act of kindness) and writing a letter of gratitude. Performing certain simple activities may improve quality of life in cancer patients and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of conducting a study of two positive activities intended to improve the psychological and interpersonal well-being of cancer patients from collectivist cultures.

SECONDARY OBJECTIVES:

I. To preliminarily assess changes in psychological, interpersonal, and physical well-being of the intervention patients and caregivers compared to control patients and caregivers.

II. To preliminarily assess changes in psychological, interpersonal, and physical well-being of patients and caregivers who are members of collectivist cultures (African American, Asian American, or Latino/Hispanic) compared to patients and caregivers who are members of individualist (European American) cultures.

EXPLORATORY OBJECTIVE:

I. To explore mechanisms through which the interventions may improve psychological and interpersonal well-being.

OUTLINE: Participants are randomized to 1 of 3 conditions.

CONDITION I (CONTRIBUTION): Patients do 1 nice thing (can be as large or as small as they wish) 2 times per week (BIW) for 4 weeks for their caregivers while at home.

CONDITION II (GRATITUDE): Patients write a letter or note of gratitude BIW for 4 weeks to their caregivers who have helped with their treatment or recovery.

CONDITION III (CONTROL): Participants keep track of their daily activities.

After completion of study, participants are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Between 35 -70 years of age
* PATIENTS: Within 1-5 years of diagnosis and actively undergoing systemic therapy, including chemotherapy, immunotherapy, endocrine and radiation therapies
* PATIENTS: Self-identify as ethnically one of the 4 ethnic groups of focus: Asian American, African American, Latino, and European American. For collectivist cultures, will aim to recruit patients of who are first- (i.e., immigrated to United States [US]) or second-generation (i.e., children of US residents who immigrated to US) immigrants
* PATIENTS: Diagnosed with any type of cancer
* PATIENTS: Able to identify a caregiver (e.g., family member) who lives in the same household, and who consents to participate in this study
* PATIENTS: Able to read, write, and speak in English
* PATIENTS: Access to internet, computer or phone, and web browser
* CAREGIVERS: Patient considers them as their caregiver
* CAREGIVERS: Lives in the same household as patient
* CAREGIVERS: Able to read, write, and speak in English
* CAREGIVERS: Access to internet, computer or phone, and web browser
* CAREGIVERS: Identifies as the same race/ethnicity group as the patient (e.g., European American wife and European American husband, or Asian American wife and Asian American husband would be pairs that are considered eligible)

Exclusion Criteria:

* PATIENTS: Life expectancy less than 6 months in the opinion of the primary physician
* PATIENTS: Inability to stand and walk on their own or with other physical limitations that preclude them from participating. (3+ on Eastern Cooperative Oncology Group [ECOG] performance status)
* PATIENTS: Major depression (e.g., as determined by a score of 10 or higher on the 10-item Center for Epidemiologic Studies Depression Scale [CES-D] at baseline, out of 30) or diagnosed prior to study (from patient records and/or self-disclosure by patient)
* CAREGIVERS: Unwilling or unable to participate in the study for any reason
* CAREGIVERS: Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Consent rate | 4 weeks
  Will calculate the 95% confidence intervals (CIs) for the consent rate.
Study completion rate | 30 days
  The study completion rate is defined as the average proportion of participants who complete follow-up assessments at the end of the study (day 30). Will also calculate the 95% CIs for the study completion rate.
Intervention adherence rate | 4 weeks
  Will calculate the 95% CIs for the intervention adherence rate.

SECONDARY OUTCOMES:
Changes in psychological well-being of the collectivist culture patients | Baseline up to 28 days
  Will calculate appropriate summary statistics and 95% CIs for the means of the Affect-Adjective Scale, Perceived Stress Scale, and Center for Epidemiologic Studies Depression Scale (CES-D) at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.
Changes in interpersonal well-being of the intervention patients | Baseline up to 28 days
  Will first calculate appropriate summary statistics and 95% CIs for the means of the Relationship Closeness Inventory at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.
Changes in physical well-being of the intervention patients | Baseline up to 28 days
  Will calculate appropriate summary statistics and 95% CIs for the means of the MD Anderson Symptom Inventory (MDASI) at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.
Changes in psychological well-being of the intervention caregivers | Baseline up to 28 days
  Will first calculate appropriate summary statistics and 95% CIs for the means of the Affect-Adjective Scale, Perceived Stress Scale, and CES-D at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.
Changes in interpersonal well-being of the intervention caregivers | Baseline up to 28 days
  Will calculate appropriate summary statistics and 95% CIs for the means of the Relationship Closeness Inventory at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.
Changes in physical well-being of the intervention caregivers | Baseline up to 28 days
  Will first calculate appropriate summary statistics and 95% CIs for the means of the MDASI at baseline, midpoint, and end of study and the outcome change score from baseline to end of study in each group.

OTHER OUTCOMES:
Potential effectiveness of the intervention | 4 weeks
  Will explore potential effects of the intervention by taking "compliance" into consideration, with compliance being defined as, e.g., completing a specified proportion of the intervention activities, so that each intervention group could be split into two or more groups based on different levels of compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shin-Cho LJ, Whisenant M, Cohen L, Chen M, Barcenas CH, Li Y, Lu Q. Feasibility, acceptability, and experienced benefits of kind acts and gratitude letter interventions among collectivist and individualist culture cancer patients and caregivers: A pilot study. Eur J Oncol Nurs. 2025 Oct;78:102970. doi: 10.1016/j.ejon.2025.102970. Epub 2025 Aug 25. PMID 40986989
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT04810052/ICF_000.pdf